CLINICAL TRIAL: NCT00002346
Title: A Phase I/II Study of Safety, Tolerance, Pharmacokinetics, and Anti-HIV Activity of 9-[2-(Bispivaloyloxymethyl)Phosphonylmethoxyethyl]Adenine (Bis-POM PMEA) and Placebo in HIV-Infected Patients
Brief Title: The Safety and Effectiveness of Bis-POM PMEA in HIV-Infected Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 232B; GS-93-402
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-03

CONDITIONS: HIV Infections
Keywords: Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents; Adenine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — adefovir dipivoxil

INTERVENTIONS:
Drug: Adefovir dipivoxil

SUMMARY:
To study the safety, tolerance, single and multiple dose pharmacokinetics, and anti-HIV activity of bis-POM PMEA ( adefovir dipivoxil ) versus placebo when administered orally on a daily basis for 2 weeks to HIV-infected patients.

DETAILED DESCRIPTION:
Patients are randomized to receive bis-POM PMEA at one of three fixed dose levels or placebo daily for 2 weeks. At each dose level, nine patients receive bis-POM PMEA and three patients receive placebo.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Prophylaxis with aerosolized pentamidine, fluconazole, ketoconazole, trimethoprim/sulfamethoxazole, or dapsone, provided a stable regimen has been maintained for at least 4 weeks prior to study entry.

Patients must have:

* HIV seropositivity.
* CD4 count >= 100 cells/mm3.
* p24 antigen (immune-complex dissociated) >= 50 pg/ml.
* Life expectancy of at least 6 months.

Prior Medication:

Allowed:

* Prior prophylaxis with aerosolized pentamidine, fluconazole, ketoconazole, trimethoprim/sulfamethoxazole, or dapsone.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active, serious infection (other than HIV infection) requiring parenteral antibiotic therapy.
* Malignancy other than cutaneous Kaposi's sarcoma.
* Clinically significant cardiac disease, including symptoms of ischemia, congestive heart failure, or arrhythmia.
* Gastrointestinal malabsorption syndrome.
* Inability to take oral medication.

Concurrent Medication:

Excluded:

* Any parenteral antibiotic therapy.
* Diuretics.
* Amphotericin B.
* Didanosine (ddI).
* Fluconazole.
* Foscarnet.
* Ganciclovir.
* Interferon-alpha.
* Interferon-beta.
* Isoniazid.
* Aminoglycoside antibiotics.
* Ketoconazole (topical allowed).
* Itraconazole.
* Rifabutin.
* Rifampin.
* Stavudine (d4T).
* Zalcitabine (ddC).
* Zidovudine (AZT).
* Lamivudine (3TC).
* Any investigational agents (except with sponsor approval).
* Systemic therapy for Kaposi's sarcoma.

Patients with the following prior condition are excluded:

History of lactose intolerance.

Prior Medication:

Excluded within 2 weeks prior to study entry:

* Any parenteral antibiotic therapy.
* Diuretics.
* Amphotericin B.
* Didanosine (ddI).
* Fluconazole.
* Foscarnet.
* Ganciclovir.
* Interferon-alpha.
* Interferon-beta.
* Isoniazid.
* Aminoglycoside antibiotics.
* Ketoconazole (topical allowed).
* Itraconazole.
* Rifabutin.
* Rifampin.
* Stavudine (d4T).
* Zalcitabine (ddC).
* Zidovudine (AZT).
* Lamivudine (3TC).
* Any investigational agents (except with sponsor approval).

Excluded within 4 weeks prior to study entry:

Systemic therapy for Kaposi's sarcoma. Active substance abuse (including alcohol) as determined by questionnaire or positive drug screen.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Univ, Baltimore, Maryland, United States

REFERENCES:
- [Background] James JS. GS 840 (adefovir dipivoxil): broad-spectrum antiviral trial, CD4 count under 100. AIDS Treat News. 1997 Feb 7;(No 264):4-5. PMID 11364103